CLINICAL TRIAL: NCT00701688
Title: Phase I Study Of The Use Of Palifermin in Pediatric Research Participants Undergoing Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Dose Escalation Study Of Palifermin in Pediatric Research Participants Undergoing Allogeneic Hematopoietic Stem Cell Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PALSCT
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-03

CONDITIONS: Oral Mucositis; Hematopoietic Stem Cell Transplantation
Keywords: Mucositis, Oral; Hematopoietic Stem Cell Transplantation; Allogeneic Transplantation; Pharmacokinetics; Maximum Tolerated Dose
MeSH Terms: conditions — Stomatitis | interventions — Fibroblast Growth Factor 7

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dose Level 1 (Experimental): Palifermin 40 mcg/kg/day intravenous
  Interventions: Drug: Palifermin
- Dose Level 2 (Experimental): Palifermin 60 mcg/kg/day intravenous
  Interventions: Drug: Palifermin
- Dose Level 3 (Experimental): Palifermin 90 mcg/kg/day intravenous
  Interventions: Drug: Palifermin

INTERVENTIONS:
Drug: Palifermin — Dose level 1 40 mcg/kg/day intravenous Dose level 2 60 mcg/kg/day intravenous Dose level 3 90 mcg/kg/day intravenous
  Other Names: Kepivance®

SUMMARY:
Mucositis is a well-known complication of both autologous and allogeneic hematopoietic stem cell transplantation (HSCT). Many who suffer this disorder require total parental nutrition and intravenous narcotics for pain control. Palifermin (Kepivance[TM]) is a human keratinocyte growth factor that is produced by recombinant DNA technology in E. coli. Palifermin is a FDA-approved, commercially available pharmacologic agent that is manufactured by Amgen. As keratinocyte growth factor receptors have been found within the epithelium of gastric mucosa, the use of palifermin has been proven to decrease the frequency and duration of severe mucositis in adult studies. Whereas the appropriate dosing regimen has been determined for adults at 60mcg/kg/day, the dosing of palifermin has not been established in the pediatric setting. This initial pediatric study of palifermin will determine the maximum tolerated dose, evaluating the use of this agent at three dose levels, below, at, and above the recommended adult dose. Non-hematologic, life-threatening NCI grade IV or grade V toxicities definitely related to the administration of palifermin from the first infusion until day +6 after HSCT (post palifermin administration day +3) will comprise the safety endpoints of the study.

The study is designed to evaluate palifermin at 3 dose levels. The study population will be recipients of either a matched family member donor or matched unrelated donor HSCT. The pharmacokinetics of palifermin at each dose level will be described to help determine the appropriate dose for future studies, which will evaluate efficacy

DETAILED DESCRIPTION:
Secondary objectives of this study include exploring the pharmacoeconomics of palifermin in this particular patient population through an assessment of inpatient days, intravenous nutrition, and analgesia requirements within 100 days post-transplantation. We will also explore the research participants' rates of immune reconstitution, specifically T and B-lymphocytes and NK cells, within the first year of HSCT.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 2 years and less than 18 years of age.
* Diagnosis of a hematologic malignancy.
* Has not received a prior autologous or allogeneic HSCT.
* Is scheduled to receive either a matched family member or MUD bone marrow stem cell graft at St. Jude Children's Research Hospital. A matched family member donor is defined as a sibling matched at 5 or 6 HLA loci or another related donor matched at 6 HLA loci.
* Is scheduled to receive a myeloablative preparative regimen (cyclophosphamide/TBI based) prior to the infusion of the allogeneic graft.
* Cardiac shortening fraction greater than or equal to 25%.
* Serum creatinine is less than twice the upper limit of normal for age.
* Bilirubin less than 3.0 mg/dl.
* Aspartate transaminase (AST) less than 500 IU/ml.
* Alanine transaminase (ALT) less than 500 IU/ml.
* Amylase less than 1.5 times the upper limits of normal for age.
* Lipase less than 1.5 times the upper limits of normal for age.
* Forced vital capacity (FVC) greater than or equal to 40% of predicted value or pulse oximetry greater than or equal to 92% on room air.
* No known hypersensitivity to E coli-derived proteins or palifermin.
* No active or recent (within 30 days prior to enrollment) gastrointestinal bleeding.
* No active or recent (within 30 days prior to enrollment) oral ulcerations.
* No active fungal infection, bacteremia or viremia within two weeks prior to enrollment.

Exclusion Criteria:

* Female - pregnant (negative serum or urine pregnancy test within 14 days prior to enrollment).
* Female - lactating.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2007-09; Primary Completion 2011-09 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose and describe the toxicity profile of palifermin in pediatric research participants with hematologic malignancies undergoing first HSCT. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Srinivasan, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org